CLINICAL TRIAL: NCT02967549
Title: Optimisation of Neonatal Ventilation - NAVA vs PAV
Brief Title: Neurally Adjusted Ventilatory Assist vs Proportional Assist Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KCH16-150
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2018-03

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAVA then PAV (Experimental): Infants randomised to NAVA then PAV
  Interventions: Device: NAVA; Device: PAV
- PAV then NAVA (Experimental): Infants randomised to PAV then NAVA
  Interventions: Device: NAVA; Device: PAV

INTERVENTIONS:
Device: NAVA — NAVA delivered by the Servo-n ventilator (Maquet)
  Other Names: neurally adjusted ventilatory assist
Device: PAV — PAV delivered by the Stephanie ventilator (Stephan)
  Other Names: Proportional Assist Ventilation

SUMMARY:
This study aims to assess whether neurally adjusted ventilatory assist or proportional assist ventilation is more effective in infants born prematurely with evolving or established bronchopulmonary dysplasia

DETAILED DESCRIPTION:
Despite improvements in survival rates of extremely preterm born infants, the incidence of bronchopulmonary dysplasia (BPD) remains unchanged over the last two decades. As invasive ventilation is frequently necessary and indeed life saving, numerous ventilator strategies have been developed to reduce damage to the developing lung. Synchronisation of mechanical breaths with the patient's respiratory effort offers the theoretical benefit of improving oxygenation and ventilation, requiring lower ventilator pressures, fewer air leaks and increased patient comfort.

Recently, novel modes of ventilation have been introduced that aim to improve upon conventional ventilation. During both proportional assist ventilation (PAV) and neurally-adjusted ventilatory assist (NAVA), respiratory support is servo-controlled based on continuous input from the baby's respiratory effort. Both aim to improve synchronization of the timing of the respiratory cycle and also to vary the level of support offered breath-to-breath in proportion to the respiratory effort of the patient.

During proportional assist ventilation (PAV), the ventilator can vary inflation pressure in phase with both volume change and flow change in order to offload both elastic and resistive components of the work of breathing. We have previously shown that PAV, compared to ACV, reduces the oxygenation index and improves respiratory muscle strength in infants born prematurely who remain ventilated at or beyond one week of life .

Neurally adjusted ventilatory assist (NAVA) utilises the electrical activity of the diaphragm to trigger the ventilator. A modified nasogastric feeding tube with a series of electrodes allows monitoring of the diaphragmatic electromyogram (Edi). The waveform of the Edi is used to trigger and control ventilator support. We have recently shown that NAVA compared to ACV results in a lower oxygenation index in infants born prematurely who remain ventilated at or beyond one week of life.

Both PAV and NAVA have been shown to have advantages above conventional triggered ventilation in neonates, but they have not been compared to each other. Our aim is to determine whether NAVA or PAV is more effective in prematurely born neonates with evolving or established BPD.

ELIGIBILITY:
Inclusion Criteria:

* Born at less than 32 weeks gestation
* ventilated at or beyond one week of life

Exclusion Criteria:

* major congenital abnormalities

Ages: 1 Week to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Oxygenation index | 2 hours
  Oxygenation index at the end of each period of ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, MD, FRCPCH, Study Director — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Background] Hunt KA, Dassios T, Greenough A. Proportional assist ventilation (PAV) versus neurally adjusted ventilator assist (NAVA): effect on oxygenation in infants with evolving or established bronchopulmonary dysplasia. Eur J Pediatr. 2020 Jun;179(6):901-908. doi: 10.1007/s00431-020-03584-w. Epub 2020 Jan 25. PMID 31980954

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02967549/Prot_SAP_000.pdf